CLINICAL TRIAL: NCT07359976
Title: Pharmacokinetic Evaluation of a Natural Hemp Extract-based Cosmetic Product After Topical and Oral Application
Brief Title: Pharmacokinetic Evaluation of a Natural CBD Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Elena Enioutina, Research Associate Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 10058347
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetics of CBD Extract, Oral and Topical Administrations
Keywords: Pharmacokinetics; CBD extract; cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral (Active Comparator)
  Interventions: Dietary Supplement: CBD extract
- Topical (Active Comparator)
  Interventions: Dietary Supplement: CBD extract

INTERVENTIONS:
Dietary Supplement: CBD extract — The purified CBD extract dissolved in the medium-chain coconut oil was administered by participants topically or orally.

SUMMARY:
The present cross-over study investigated whether cannabidiol (CBD) or its metabolites and delta-9-tetrahydrocannabinol (THC) can be detected in the systemic circulation following a single topical application of a natural hemp extract-based cosmetic (NHEC) consisting of CBD and medium chain triglycerides (capric, caprylic triglycerides or medium chain triglycerides (MCT)) derived from coconut oil. Since consumers can consider hemp/CBD oil as a nutritional product or dietary supplement, it can be ingested by consumers. Therefore, we analyzed the concentrations of CBD, THC, and their metabolites in systemic circulation after oral NHEC administration. Additionally, we tested whether a single topical or oral use of the NHEC would lead to detectable levels of THC in the urine samples using Easy@Home THC detection strips. This study has no intent to treat or prevent any diseases or conditions.

In this study, volunteer participants were assigned to one of two study groups: Cohort A (oral administration) or Cohort B (topical administration). After completing the study in the first assigned Cohort, participants had a 15-day washout period before beginning the study in the next Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers (males and females, 18 - 50 years old) with a BMI 19-30. Subjects who were able to ingest or apply test products. The participants understood the requirements of the study.

Exclusion Criteria:

1. Individuals less than 18 years of age or over 50 years of age at enrollment;
2. Individuals previously participated in a research study involving administration of the investigational compound within one month prior to the current study;
3. Individuals who were using any recreational drug, specifically marijuana, in the past six months;
4. Individuals with a history of alcoholism;
5. Individuals who have conditions that might have possible interference with the study product absorption, distribution, metabolism, or excretion: previous surgery of the gastrointestinal tract, including removal of parts of the stomach, bowel, liver, gall bladder, pancreas or adjustable gastric band surgery, impaired glucose tolerance, diabetes mellitus, renal disease, edema, hepatic disorder.
6. Individuals who are pregnant or may become pregnant during studies
7. Individuals who are reporting any chronic diseases, such as mental disorders
8. The University of Utah faculty, students, and employees whom the investigators of this study directly supervise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Analysis of CBD, THC, and their metabolites in the plasma of participants | 24 hours
  Since the general consumers may use oil-based CBD extract as topical cream or as a dietary supplement, this crossover study intended to characterizes the PK of the concentrations of CBD, THC, and their metabolites in the plasma of healthy volunteers receiving a single topical or oral dose of a natural hemp extract-based cosmetic (NHEC) consisting of CBD and medium-chain triglycerides (MTC) derived from coconut oil.

SECONDARY OUTCOMES:
Urine THC | 24 hours
  Since the general public reports positive urine THC tests when using CBD oils, to determine whether the participants who used NHEC would have positive urine THC tests.
Bioavalability | 24 hours
  To calculate the bioavailability of NHEC following topical or oral administrations using the published bioavailability data

CONTACTS AND LOCATIONS:
Locations (1):
- Division Clinical Pharmacology, SOM, University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No